CLINICAL TRIAL: NCT03229811
Title: Integrating Conservative Kidney Management Options and Advance Care Planning Into a Pre-Dialysis Educational Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI left academic practice
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nwamaka Eneanya, MD, MPH, Attending Nephrologist, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 831500
Record Dates: First submitted 2017-07-21; First posted 2017-07-26 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Advance Care Planning; Chronic Kidney Diseases; Conservative Kidney Management
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Comprehensive pre-dialysis program incorporating conservative and advance care planning education
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pre-dialysis education (No Intervention): Standard pre-dialysis options education including hemodialysis, peritoneal dialysis, and kidney transplantation
- ESRD education + ACP (Active Comparator): Standard ESRD education + conservative kidney management and advance care planning education
  Interventions: Other: ESRD education + conservative kidney management and ACP education

INTERVENTIONS:
Other: ESRD education + conservative kidney management and ACP education — Targeted conservative kidney management and advance care planning education delivered in person by trained healthcare providers
  Arms: ESRD education + ACP

SUMMARY:
The goals of this work will be to evaluate the preliminary efficacy of a comprehensive pre-dialysis education program on increased knowledge of conservative kidney management and advance care planning among patients with advanced CKD.

DETAILED DESCRIPTION:
This intervention will be randomized among patients with advanced chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Stage 4 or 5 CKD (defined by the CKD-EPI estimation of GFR < 30 ml/min/1.73m2)
* Age 65 years or greater or frail
* self-reported Black or White race

Exclusion Criteria:

* History of dementia
* History of legal blindness
* Listed for kidney transplantation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stallings TL, Temel JS, Klaiman TA, Paasche-Orlow MK, Alegria M, O'Hare A, O'Connor N, Dember LM, Halpern SD, Eneanya ND. Integrating Conservative kidney management Options and advance care Planning Education (COPE) into routine CKD care: a protocol for a pilot randomised controlled trial. BMJ Open. 2021 Feb 22;11(2):e042620. doi: 10.1136/bmjopen-2020-042620. PMID 33619188

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Pre-dialysis Education | ESRD Education + ACP
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 4 enrolled participants were randomized to the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Pre-dialysis Education | ESRD Education + ACP | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 76 (6.06) | 76 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 4 | 4
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 2 | 2
  White |  | 2 | 2
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Conservative Kidney Management and Advance Care Planning (Pre-intervention)
Description: Knowledge of conservative kidney management and advance care planning pre-intervention (mean score) Total score ranges from 0 to 9, where 9 represents having the most knowledge about conservative kidney management and advance care planning
Time Frame: Pre-intervention and Day 1 post-intervention
Population: No participants were randomized to standard education
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Pre-dialysis Education | ESRD Education + ACP
Number analyzed (Participants) | 0 | 4
score on a scale |  | 5.75 (3.60)

2. Primary Outcome: Knowledge of Conservative Kidney Management and Advance Care Planning (Post-intervention)
Description: Knowledge of conservative kidney management and advance care planning post-intervention (mean score) Total score ranges from 0 to 9, where 9 represents having the most knowledge about conservative kidney management and advance care planning
Time Frame: Immediate post-intervention
Population: No participants were randomized to standard education. One enrolled participant did not complete the post-knowledge questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Pre-dialysis Education | ESRD Education + ACP
Number analyzed (Participants) | 0 | 3
score on a scale |  | 8.67 (0.58)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 month
Description: All-Cause Mortality were not monitored/assessed
Arm/Group | Standard Pre-dialysis Education | ESRD Education + ACP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
This trial was terminated early leading to a small number of participants who where analyzed. Data should be interpreted cautiously given this caveat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT03229811/Prot_SAP_000.pdf